CLINICAL TRIAL: NCT01837121
Title: a Randomized Controlled Trail to Determine the Impact of a SMS Reminder Among Diabetic Retinopathy Patients in Rural China
Brief Title: a Trial of Using SMS Reminder Among Diabetic Retinopathy Patients in Rural China
Acronym: SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Orbis (Other); The World Diabetes Foundation (Other)
Responsible Party: Principal Investigator, Congdon Nathan, vice director,Blindness Prevention and Treatment Department, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ZOC-WDF-SMS
Record Dates: First submitted 2013-04-14; First posted 2013-04-22 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Compliance; Diabetic Retinopathy; SMS
Keywords: not-attended rate; re-visit; vision; knowledge; satisfaction
MeSH Terms: conditions — Patient Compliance; Diabetic Retinopathy; Personal Satisfaction

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the SMS group (Other): the diabetic retinopathy patient in the SMS group will receive a SMS reminder message about the revisit time,address 1 week and 3 day before the appointment.
  Interventions: Other: the SMS reminder message
- the control group (No Intervention): the diabetic retinopathy patient in the control group won't get any reminder message before the appointment.

INTERVENTIONS:
Other: the SMS reminder message — the SMS reminder message will sent to the SMS group patients 1 week and 3 day before there appointment,to remind them the exact time and address of the revisit appointment.
  Arms: the SMS group

SUMMARY:
The purpose of this study is to use a randomized controlled design to determine the impact of a SMS messaging intervention on the following outcomes among persons diagnosed with diabetic retinopathy in rural China.

DETAILED DESCRIPTION:
SMS message reminder is a system which can sent re-visit information to remind the patient about the revisit time and address. The investigators can use the SMS system to find out if it is a useful to reduce the not-attended rate of the revisit appointment among the rural diabetic retinopathy patients.

ELIGIBILITY:
Inclusion Criteria:

- all the diabetes patients who would like to join our study in 5 CREST cooperated rural hospitals.

Exclusion Criteria:

1. Both the patient and his/her caretakers don't have cellphone,or the one who has cellphone but don't know how to use the SMS function.
2. The first re-visit appointment time is outside our study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Not-attended rate | up to 1.5 years
  Compare the SMS patient not-attended rate with the control group to show the impact of SMS reminder on the compliance with scheduled follow-up visit

SECONDARY OUTCOMES:
Knowledge about Diabetic retinopathy on a standardized examination | up to 1.5 years
  Using a questionnaire about the comprehensive eye exam and Diabetic retinopathy to compare Knowledge about Diabetic retinopathy on a standardized examination between the SMS group and the control group
Presenting vision | up to 1.5 years
  Presenting vision(Best corrected visual acuity) in the better-seeing and worse-seeing eyes of the two group
Loss of presenting vision | up to 1.5 years
  Loss of presenting vision(Best corrected visual acuity) in better-seeing eye thought due to Diabetic retinopathy
Satisfaction with care | up tp 1.5 years
  Using a patient satisfaction questionnaire to compare satisfaction with care between the SMS group and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Nathan G Congdon, MD,MPH, Study Director — Blindness Prevention and Treament Department,Zhongshan Ophthalmic Center
Locations (1):
- Blindness Preventment and Treatment Department, Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China